CLINICAL TRIAL: NCT02564224
Title: Randomized Clinical Trial of Stoma Reversal Comparing Pursestring Wound Closure vs Conventional Closure to Eliminate the VSS Score of the Scar for Colorectal Cancer Patients
Brief Title: Study Comparing Pursestring Wound Closure vs Conventional Closure to Reverse Stoma of Colorectal Cancer Patients
Acronym: PURSE
Status: No longer available | Type: Expanded Access
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, the Second Affiliated Hospital of Zhejiang University, Zhejiang University
Other Study IDs: CRCCZ-S01
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Colorectal Cancer; Stoma Closure Technic
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Procedure: Pursestring Wound Closure — Procedure: Pursestring Wound Closure
Procedure: Conventional Wound Closure — Procedure: Conventional Wound Closure
Device: prolene

SUMMARY:
Temporary stomas has been performed to reduce complications after colorectal cancer surgery, especially in high-risk anastomosis. Different closure technics showed different outcome. The aim of this study is to compare the scar length , surgical site infection and pain score of purse-string wound closure vs conventional closure.

ELIGIBILITY:
Inclusion Criteria:

* Receiving temporary ostomy because of colorectal cancer at least 3 months ago;
* Age of≥18 and ≤80

Exclusion Criteria:

* Not willing or incapable to comply with all study visits and assessments
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that puts the patient at high risk for treatment-related complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang, China